CLINICAL TRIAL: NCT04654078
Title: An Open-label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics and Safety of IN-C004 in Healthy Volunteers
Brief Title: Study to Evaluate the Pharmacokinetic Characteristics and Safety of IN-C004 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_KOD_102
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Group 1
  Interventions: Drug: IN-C004 with water; Drug: IN-C004 without water; Drug: K-CAB tab. with water
- Group 2 (Experimental): Group 2
  Interventions: Drug: IN-C004 with water; Drug: IN-C004 without water; Drug: K-CAB tab. with water
- Group 3 (Experimental): Group 3
  Interventions: Drug: IN-C004 with water; Drug: IN-C004 without water; Drug: K-CAB tab. with water
- Group 4 (Experimental): Group 4
  Interventions: Drug: IN-C004 with water; Drug: IN-C004 without water; Drug: K-CAB tab. with water
- Group 5 (Experimental): Group 5
  Interventions: Drug: IN-C004 with water; Drug: IN-C004 without water; Drug: K-CAB tab. with water
- Group 6 (Experimental): Group 6
  Interventions: Drug: IN-C004 with water; Drug: IN-C004 without water; Drug: K-CAB tab. with water

INTERVENTIONS:
Drug: IN-C004 with water — One time dose of IN-C004 taken with water
  Other Names: IN-C004
Drug: IN-C004 without water — One time dose of IN-C004 taken without water
  Other Names: IN-C004
Drug: K-CAB tab. with water — One time dose of K-CAB tab. taken with water
  Other Names: K-CAB tab.

SUMMARY:
To evaluate the pharmacokinetic characteristics and safety of IN-C004 in healthy volunteers

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose, Crossover Study

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥19.0 kg/m2 and ≤27.0 kg/m2 with a body weight ≥ 45 kg at screening.

Exclusion Criteria:

* History or evidence of clinically significant disease
* History of drug/alcohol abuse
* Participated in other studies and received investigational products within 6 months prior to the first study dose.
* AST(GOT) or ALT(GPT) > 2 X upper limit of normal at screening
* Not able to use a medically acceptable contraceptive method throughout the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
AUCt of tegoprazan | pre-dose(0 hour), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Area under the plasma concentration-time curve of tegoprazan
Cmax of tegoprazan | pre-dose(0 hour), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Maximum Plasma Concentration at Steady State of tegoprazan
AUCt of tegoprazan metabolite M1 | pre-dose(0 hour), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hour
  Area under the plasma concentration-time curve of tegoprazan metabolite M1
Cmax of tegoprazan metabolite M1 | pre-dose(0 hour), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours
  Maximum Plasma Concentration at Steady State of tegoprazan metabolite M1

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea